CLINICAL TRIAL: NCT01585441
Title: Phase II, Randomized, Placebo-Controlled Study for the Evaluation of Finasteride in the Treatment of Chronic Central Serous Chorioretinopathy
Brief Title: Finasteride for Chronic Central Serous Chorioretinopathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated early due to lack of enrollment.
Sponsor: National Eye Institute (NEI) (NIH)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 120119; 12-EI-0119
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-11

CONDITIONS: Retinal Disease
Keywords: Finasteride; Central Serous Chorioretinopathy
MeSH Terms: conditions — Retinal Diseases; Central Serous Chorioretinopathy | interventions — Finasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Finasteride 5 mg (Experimental): Participants randomly assigned to the finasteride 5 mg arm were instructed to take one capsule daily for three months.
  Interventions: Drug: Finasteride
- Placebo (Placebo Comparator): Participants randomly assigned to the placebo arm will instructed to take one capsule daily for three months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Finasteride — Finasteride is available as white, round 5 mg tablets. During the masked period, the tablets are re-formulated in capsules with inactive ingredients. The re-formulated finasteride capsules are indistinguishable from the placebo capsules.
  Other Names: Propecia®; Proscar®
  Arms: Finasteride 5 mg
Drug: Placebo — Capsule with no active ingredients to mimic finasteride
  Arms: Placebo

SUMMARY:
Background:

* Central serous chorioretinopathy (CSC) is a disease that causes fluid to collect under the retina. It affects the macula, which is in the center of the retina and is needed for sharp, clear vision. In many cases, CSC resolves on its own and does not need treatment. However, in some cases it does not go away or comes back after treatment. This is known as chronic CSC.
* Chronic CSC may be caused by hormones called androgens. Finasteride is a drug that can alter the effects certain of androgens. Researchers want to compare finasteride with a placebo to see if it is a safe and effective treatment for chronic CSC.

Objectives:

- To see if finasteride is a safe and effective treatment for chronic CSC.

Eligibility:

- Individuals at least 18 years of age who have chronic CSC in one or both eyes.

Design:

* Participants will be screened with a physical exam and medical history. A full eye exam will be performed. Blood and urine samples will also be collected.
* Some participants may have photodynamic therapy (PDT), the standard treatment for CSC. PDT helps to reduce the amount of fluid in the eye. Participants will need to wait for 3 months after PDT before starting the finasteride study.
* Participants will be separated into two groups. One group will take finasteride 5 mg (formulated into capsules); the other group will take a placebo capsule. All participants will take the capsules for 3 months.
* After 3 months on the assigned capsule (finasteride or placebo), all participants will have the opportunity to take finasteride for at least another 4 years and 9 months. This phase of the study is optional.
* Participants will have regular study visits. At each visit, they will have physical exams and eye exams. They will also provide blood and urine samples.
* During the first 3 months, participants will have 2 study visits. After 3 months, if the participant continues in the optional (or as needed) phase of the protocol, visits will occur at Month 6, Month 12 and every 12 months thereafter. However, additional visits may be needed.

DETAILED DESCRIPTION:
Objective:

Central serous chorioretinopathy (CSC) is a chorioretinal disorder characterized by an accumulation of serous fluid under the retina. Although acute CSC tends to resolve spontaneously on its own with minimal sequelae, chronic CSC tends to persist and lead to irreversible visual loss. The pathogenesis of CSC is complex. However, systemic androgens have been implicated. Finasteride is an anti-androgen medication that is widely used in the treatment of various conditions. A previous study performed at the NEI demonstrated a reduction in the amount of subretinal fluid among participants treated with 5 mg of finasteride. The objective of this study is to further investigate the efficacy of oral finasteride as a treatment for chronic CSC.

Study Population:

Thirty-eight participants with chronic CSC are eligible. Up to an additional four participants may be enrolled to account for participants who withdraw from the study prior to Month 3.

Design:

In this Phase II, single-center, placebo-controlled, double-masked, randomized trial, investigational product will be administered to two different groups. Half of the participants will be randomized to 5 mg oral finasteride for the initial three months. The other half of the participants will be randomized to placebo for the first three months. At the end of three months of treatment, all participants may be followed for at least four years and nine months. During this follow-up period, all participants will be able to receive finasteride therapy pro re nata (PRN) if subretinal fluid re-emerges. The PRN phase will last until the last participant completes the five years of follow-up. Other standard care treatments, such as photodynamic therapy, will also be permitted after the primary outcome at three months.

Outcome Measures:

The primary outcome for regulatory filing is the proportion of participants with an improvement in best-corrected visual acuity (BCVA) ≥ 15 letters at three months compared to baseline in the study eye. The primary outcome for publication of the study results is the proportion of participants with a subretinal fluid volume decrease ≥ 50% at three months compared to baseline in the study eye. Secondary efficacy outcomes include changes in BCVA, changes in the maximum retinal volume as measured on optical coherence tomography (OCT), changes in central retinal thickness on OCT, changes in leakage as seen on fluorescein angiography (FA), changes in size of existing plaque(s) on indocyanine green (ICG) angiography, changes in autofluorescence patterns seen on fundus autofluorescence (FAF) imaging, changes in mean macular sensitivity as assessed by microperimetry, changes in serum levels of testosterone and dihydrotestosterone (DHT), as well as changes in urine levels of cortisol during the study period. Safety outcomes include the number and severity of adverse reactions from the investigational product and the number of withdrawals.

ELIGIBILITY:
INCLUSION CRITERIA:

* Participant must have chronic Central Serous Chorioretinopathy (CSC) in at least one eye as defined by all of the following criteria. This eye will be referred to as the study eye.
* The presence of subretinal fluid, as determined by optical coherence tomography (OCT), AND
* The subretinal fluid must have been present for at least three months or recurrent in cases of chronic CSC/diffuse retinal pigment epitheliopathy, AND/OR
* The presence of characteristic fluorescein angiographic or autofluorescence features of CSC, such as one or more pinpoint leaks and/or diffuse retinal pigment epitheliopathy noted on fluorescein or descending tract lesions on autofluorescence.
* Participant must have a steady fixation in the study eye.
* Participant must have media clear enough in the foveal or parafoveal area in the study eye for good quality photographs.
* Participant must have visual acuity between 20/25 and 20/400 in the study eye.

EXCLUSION CRITERIA:

* Participant has evidence of choroidal neovascularization (CNV) in the study eye.
* Participant is expected to need ocular surgery in the study eye during the first three months of the study.
* Participant has had photodynamic therapy (PDT) or focal laser treatment in the study eye within three months prior to enrollment or is expected to need PDT or focal laser treatment in the study eye during the first three months of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Y Chew, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gomolin JE. Choroidal neovascularization and central serous chorioretinopathy. Can J Ophthalmol. 1989 Feb;24(1):20-3. PMID 2469527
- [Background] Tewari HK, Gadia R, Kumar D, Venkatesh P, Garg SP. Sympathetic-parasympathetic activity and reactivity in central serous chorioretinopathy: a case-control study. Invest Ophthalmol Vis Sci. 2006 Aug;47(8):3474-8. doi: 10.1167/iovs.05-1246. PMID 16877418
- [Background] Spahn C, Wiek J, Burger T, Hansen L. Psychosomatic aspects in patients with central serous chorioretinopathy. Br J Ophthalmol. 2003 Jun;87(6):704-8. doi: 10.1136/bjo.87.6.704. PMID 12770965
- [Derived] Lange CA, Qureshi R, Pauleikhoff L. Interventions for central serous chorioretinopathy: a network meta-analysis. Cochrane Database Syst Rev. 2025 Jun 16;6(6):CD011841. doi: 10.1002/14651858.CD011841.pub3. PMID 40522203

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Finasteride 5 mg | Placebo
Started | 3 | 3
Month 3 | 2 (One participant was not evaluated at Month 3 but at the final visit due to study terminating early.) | 3
Received Finasteride at Month 3 | 2 | 2
Final Study Safety Visit | 3 | 2 (A final study visit was not required for the placebo participant who completed the study at Month 3.)
Completed | 3 (Defined as completing the Month 3 masked phase of the study and/or the final safety visit) | 3 (Defined as completing the Month 3 masked phase of the study and/or the final safety visit)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Finasteride 5 mg | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With an Improvement in Best-corrected Visual Acuity (BCVA) ≥ 15 Letters at 3 Months Compared to Baseline.
Description: This is the regulatory filing primary outcome measure. Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20.
Time Frame: Month 3
Measure: Number; unit: participants
Units Other Than Participants: Eyes
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 2 | 3
Number analyzed (Eyes) | 2 | 3
participants | 0 | 0

2. Primary Outcome: Proportion of Participants With a Reduction in Subretinal Fluid Volume ≥ 50% at 3 Months Compared to Baseline
Description: This is the primary outcome measure for publication of study results. Subretinal fluid volume will be determined by manually moving the segmentation lines of the optical coherence tomography (OCT) image using the "Edit Segmentation" function of the Cirrus™ HD-OCT software. The segmentation lines will be edited to outline the inner and outer borders of the subretinal fluid pocket. This will be done manually for all the individual B-scans of each OCT image, after which the software algorithm automatically calculates the subretinal fluid volume.
Time Frame: Month 3
Measure: Number; unit: participants
Units Other Than Participants: Eyes
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 2 | 3
Number analyzed (Eyes) | 2 | 3
participants | 1 | 0

3. Secondary Outcome: Number of Participants With Adverse Reactions Related to the Investigational Product
Description: The outcome measure refers only to events that were classified as related to the investigational product.
Time Frame: Duration of the study, up to 1.5 years
Measure: Number; unit: participants
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 3 | 3
participants | 0 | 1

4. Secondary Outcome: Number of Participants Who Withdrew From the Study
Time Frame: Duration of the study, up to 1.5 years
Measure: Number; unit: participants
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 3 | 3
participants | 0 | 0

5. Secondary Outcome: Changes in Best-corrected Visual Acuity (BCVA) in the Study Eye at Month 3 Compared to Baseline
Description: Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20.
  A positive change value indicates improvement of the outcome. A negative change value indicates worsening of the outcome.
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: Eyes
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 2 | 3
Number analyzed (Eyes) | 2 | 3
ETDRS letters | 1.00 (1.41) | 1.67 (2.08)

6. Secondary Outcome: Changes in Best-corrected Visual Acuity (BCVA) in the Study Eye at the Safety Visit Compared to Baseline
Description: as for outcome 5
Time Frame: Final Study Visit
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: Eyes
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 3 | 2
Number analyzed (Eyes) | 3 | 2
ETDRS letters | -3.33 (8.39) | 0.50 (0.71)

7. Secondary Outcome: Percent Change in Subretinal Fluid Volume in the Study Eye at Month 3 Compared to Baseline
Description: Subretinal fluid volume will be determined by manually moving the segmentation lines of the optical coherence tomography (OCT) image using the "Edit Segmentation" function of the Cirrus™ HD-OCT software. The segmentation lines will be edited to outline the inner and outer borders of the subretinal fluid pocket. This will be done manually for all the individual B-scans of each OCT image, after which the software algorithm automatically calculates the subretinal fluid volume.
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: percent change
Units Other Than Participants: Eyes
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 2 | 3
Number analyzed (Eyes) | 2 | 3
percent change | -37.50 (53.03) | 27.78 (63.10)

8. Secondary Outcome: Changes in Mean Macular Sensitivity in the Study Eye at Month 3 Compared to Baseline
Description: Microperimetry was used to assess macular sensitivity.
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: decibels
Units Other Than Participants: Eyes
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 2 | 3
Number analyzed (Eyes) | 2 | 3
decibels | -2.00 (3.82) | -1.40 (1.47)

9. Secondary Outcome: Changes in Mean Macular Sensitivity in the Study Eye at the Safety Visit Compared to Baseline
Description: Microperimetry was used to assess macular sensitivity.
Time Frame: Final Study Visit
Measure: Mean (Standard Deviation); unit: decibels
Units Other Than Participants: Eyes
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 3 | 2
Number analyzed (Eyes) | 3 | 2
decibels | -2.03 (3.91) | -2.45 (0.50)

10. Secondary Outcome: Change in Central Retinal Thickness in the Study Eye at Month 3 Compared to Baseline
Description: Central retinal thickness was assessed by spectral-domain optical coherence tomography (SD-OCT).
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: μm
Units Other Than Participants: Eyes
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 2 | 3
Number analyzed (Eyes) | 2 | 3
μm | -55.00 (50.91) | 20.33 (72.59)

11. Secondary Outcome: Change in Central Retinal Thickness in the Study Eye at the Safety Visit Compared to Baseline
Description: Central retinal thickness was assessed by spectral-domain optical coherence tomography (SD-OCT).
Time Frame: Final Study Visit
Measure: Mean (Standard Deviation); unit: μm
Units Other Than Participants: Eyes
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 3 | 2
Number analyzed (Eyes) | 3 | 2
μm | -39.67 (93.30) | 50.50 (41.72)

12. Secondary Outcome: Change in Serum Dihydrotestosterone (DHT) Concentration at Month 3 Compared to Baseline
Description: The mean change is reported in picograms of DHT per milliliter of serum.
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 2 | 3
pg/mL | -332.00 (176.78) | -93.67 (113.50)

13. Secondary Outcome: Change in Serum Dihydrotestosterone (DHT) Concentration at the Safety Visit Compared to Baseline
Description: The mean change is reported in picograms of DHT per milliliter of serum.
Time Frame: Final Study Visit
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 3 | 2
pg/mL | -101.67 (103.00) | -337.50 (467.40)

14. Secondary Outcome: Change in Serum Testosterone Concentration at Month 3 Compared to Baseline
Description: The mean change is reported in nanograms of testosterone per decaliter of serum.
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 2 | 3
ng/dL | -33.50 (139.30) | -29.67 (111.96)

15. Secondary Outcome: Change in Serum Testosterone Concentration at the Safety Visit Compared to Baseline
Description: The mean change is reported in nanograms of testosterone per decaliter of serum.
Time Frame: Final Study Visit
Measure: Mean (Standard Deviation); unit: ng/dL
Units Other Than Participants: Eyes
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 3 | 2
Number analyzed (Eyes) | 3 | 2
ng/dL | -42.00 (194.51) | 33.00 (100.41)

16. Secondary Outcome: Change in Urinary Levels of Cortisol at Month 3 Compared to Baseline
Description: The mean change is reported in micrograms (μg).
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: μg
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 2 | 3
μg | 5.75 (23.12) | -7.10 (16.71)

17. Secondary Outcome: Change in Urinary Levels of Cortisol at the Safety Visit Compared to Baseline
Description: The mean change is reported in micrograms (μg).
Time Frame: Final Study Visit
Population: One finasteride participant's cortisol lab value could not be calculated due to Cortisol, Urine <1.5 ng/mL.
Measure: Mean (Standard Deviation); unit: μg
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 2 | 2
μg | -0.60 (3.53) | 0.70 (6.08)

18. Secondary Outcome: Number of Participants Presenting No Change in Autofluorescence Patterns at Month 3 Compared to Baseline
Description: Autofluorescence patterns as observed on Fundus Autofluorescence (FAF) imaging
Time Frame: Month 3
Measure: Number; unit: participants
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 2 | 3
participants | 2 | 3

19. Secondary Outcome: Number of Participants Presenting No Change in Autofluorescence Patterns at the Safety Visit Compared to Baseline
Description: Autofluorescence patterns as observed on Fundus Autofluorescence (FAF) imaging
Time Frame: Final Study Visit
Population: One placebo participant was not evaluated at the final safety visit, as the participant completed the study at the Month 3 visit.
Measure: Number; unit: participants
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 3 | 2
participants | 3 | 2

20. Secondary Outcome: Number of Participants Presenting No Change in Size of Existing Plaque(s) on Indocyanine Green (ICG) Angiography at Month 3 Compared to Baseline
Time Frame: Month 3
Measure: Number; unit: participants
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 2 | 3
participants | 2 | 3

21. Secondary Outcome: Number of Participants Presenting No Change in Size of Existing Plaque(s) on Indocyanine Green (ICG) Angiography at the Safety Visit Compared to Baseline
Time Frame: Final Study Visit
Population: as for outcome 19
Measure: Number; unit: participants
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 3 | 2
participants | 3 | 2

22. Secondary Outcome: Number of Participants Presenting No Change in Fluid Leakage at Month 3 Compared to Baseline
Description: Changes in leakage as observed on fluorescein angiography (FA)
Time Frame: Month 3
Measure: Number; unit: participants
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 2 | 3
participants | 2 | 2

23. Secondary Outcome: Number of Participants Presenting No Change in Fluid Leakage at the Safety Visit Compared to Baseline
Description: Changes in leakage as observed on fluorescein angiography (FA)
Time Frame: Final Study Visit
Measure: Number; unit: participants
Arm/Group | Finasteride 5 mg | Placebo
Number analyzed (Participants) | 3 | 2
participants | 2 | 2

ADVERSE EVENTS:
Time Frame: Duration of the study, up to 1.5 years
Arm/Group | Finasteride 5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 2/3 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Finasteride 5 mg (N=3) | Placebo (N=3)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Eye pruritis (Eye disorders) | 1 (1) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated early due to lack of enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes